CLINICAL TRIAL: NCT05460650
Title: Evaluation of Acceptance and Usability of an App Promoting Healthy Behaviours Amongst Young Women at Increased Risk of Breast Cancer
Brief Title: Acceptance and Usability of an App Promoting Healthy Behaviours Amongst Young Women at Increased Risk of Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Mary Pegington, Senior Research Dietitian, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REC 22/WA/0164
Record Dates: First submitted 2022-06-23; First posted 2022-07-15 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer; Overweight and Obesity; Diet, Healthy; Weight Gain; Alcohol Drinking; Smoking Behaviors; Healthy Nutrition; Healthy Lifestyle; Healthy Eating Index
MeSH Terms: conditions — Breast Neoplasms; Overweight; Obesity; Weight Gain; Alcohol Drinking; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Receives app (Experimental): All women in the study will receive access to the app.
  Interventions: Behavioral: App Promoting Healthy Behaviours

INTERVENTIONS:
Behavioral: App Promoting Healthy Behaviours — Women on the study will receive two months access to the app.

SUMMARY:
It is estimated that around 20% of breast cancers (BC) in the UK are preventable through adherence to appropriate health behaviours, i.e., healthy diet, physical activity, limited alcohol, not smoking, and that women at increased risk of BC could benefit from greater decreases in risk than the general population via health behaviour changes. Young women (age <35 years) who are at increased risk of developing BC currently receive little or no information regarding health behaviours and BC risk, or support for behaviour change. This feasibility study aims to explore whether a novel app is acceptable to women at increased risk and could potentially engage them with improved health behaviours which could reduce their future risk of BC.

DETAILED DESCRIPTION:
Aims

1. To assess the acceptability and usability of the app to young women at increased risk of BC
2. To assess the feasibility of study procedures before running a future efficacy study using the app as an intervention

Objectives

1. Explore views of users of the experiences during and after using the app
2. Explore views of users on their experience of the two different recruitment procedures (targeted mailshot, or social media, newsletters and websites), and the online consent procedure.
3. Interpret user data from the app including frequency and patterns of use of the different functions
4. Analyse recruitment data to explore how the two different recruitment procedures could be improved for the next study
5. Assemble a list of suggested changes to recruitment and consent procedures, and to the app, to be considered before the next study.
6. Quantify health care professional (HCP) time required for administering the private Facebook chat group, and through e-mail/private message support.
7. Quantify researcher time required for cleaning and analysis of app data.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-35 years
* Live in the UK
* Moderate or high risk of BC (see 6.5 for definition)
* Ability to communicate in English
* Ability to download and use an app (available on both ioS and Android)

Exclusion Criteria:

* Previous BC (other cancers will not be excluded)
* Previous preventative mastectomy
* Currently trying to gain weight
* Previous weight loss surgery
* Currently taking weight loss medication, prescribed (for example orlistat, liraglutide, Naltrexone/Bupropion [Mysimba]) or other
* Have a medical condition that influences diet and weight, for example, diabetes, inflammatory bowel disease or cystic fibrosis
* Current diagnosis of a psychiatric disorder, for example bipolar psychotic disorder or current self-harm
* Current alcohol or drug dependency
* Current or previous diagnosis of an eating disorder

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Acceptability and usability of the app | Two months
  Assess acceptability and usability of the app by interviews

SECONDARY OUTCOMES:
Acceptability of study recruitment, consent and trial procedures | Two months
  Assess the feasibility of all study procedures by interviews by thematic analysis of transcripts
Study uptake numbers via invite letter and social media posts | Two months
  Recruitment source of the participants from recruitment data, e.g. percentage response to mailshot, percentage uptake, number recruited via the postal invite letter and via social media
Acceptability and usability of the app via questionnaire | Two months
  Acceptability of the app, barriers and facilitators to engagement, likes and don't likes within app, usability, likelihood of extended use via questionnaire.
Errors in app data entry | Two months
  Quantification of errors in information inputted by participants, e.g. kg entered as stones and pounds.
Number of interactions with the private Facebook group | Two months
  Number of participant interactions in the Facebook group during the two months.

CONTACTS AND LOCATIONS:
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
After data analysis is complete, the fully anonymised data will be uploaded on to Figshare as per University of Manchester guidance and will remain there indefinitely.
Supporting Information: Study Protocol, SAP
Time Frame: After data analysis is complete, the fully anonymised data will be uploaded on to Figshare as per University of Manchester guidance and will remain there indefinitely.

REFERENCES:
- [Derived] Pegington M, Davies A, Mueller J, Cholerton R, Howell A, Evans DG, Howell SJ, French DP, Harvie M. Evaluating the Acceptance and Usability of an App Promoting Weight Gain Prevention and Healthy Behaviors Among Young Women With a Family History of Breast Cancer: Protocol for an Observational Study. JMIR Res Protoc. 2022 Dec 16;11(12):e41246. doi: 10.2196/41246. PMID 36525287

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-26): https://cdn.clinicaltrials.gov/large-docs/50/NCT05460650/Prot_SAP_000.pdf